CLINICAL TRIAL: NCT04379661
Title: SUNLIGHT Study: Online Support Groups for Multiple Sclerosis (MS) to Address COVID-19
Brief Title: SUNLIGHT Study: Online Support Groups for MS to Address COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Victoria M. Leavitt, Assistant Professor of Neuropsychology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS9939
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: MS (Multiple Sclerosis); COVID-19; Support Groups
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online support group (Experimental): Online weekly 1-hour moderated support group sessions for 12-weeks; participants complete surveys at baseline and 12-week follow-up
  Interventions: Behavioral: Online support Group
- Treatment as usual (No Intervention): Inactive control group of participants who complete surveys at baseline and 12-weeks later

INTERVENTIONS:
Behavioral: Online support Group — 12 one-hour, once-weekly online support groups for people with Multiple Sclerosis to address anxiety related to the COVID-19 outbreak and its effects on them.
  Arms: Online support group

SUMMARY:
Stress and anxiety can have an adverse impact on health, and the experience of many around the 2020 outbreak of COVID-19 is affecting health and well-being. Individuals with chronic disease such as multiple sclerosis may be particularly vulnerable in some ways, but also particularly resilient in others. This study evaluates the effects of belonging to online support groups that meet weekly for 12 weeks to address the stress and anxiety felt by individuals with Multiple Sclerosis (MS). This study will also measure and explore the effects of online support groups.

DETAILED DESCRIPTION:
Anxiety is a pervasive and debilitating symptom for individuals with MS, who are at much greater risk for anxiety than the general population. The lifetime prevalence of anxiety in MS is estimated at 48.9%, compared to 37.9% in the general population. The negative consequences of anxiety for individuals with MS include impairment of work function and workplace attrition, increased healthcare usage and healthcare costs, increased physical disability (i.e., higher Expanded Disability Status Scale (EDSS) score), and reduced overall quality of life. And while anxiety has been shown to be acutely elevated both before and in the first years after diagnosis, individuals with longstanding MS also exhibit anxiety at higher rates than the general population. Of note, women are at heightened risk for both anxiety and MS, and lower socioeconomic status (SES) is associated with increased prevalence of anxiety in MS. In the SUNLIGHT study, participants join a structured meeting in which they receive content specifically focused on anxiety, its detrimental impact on individuals with MS, and an emphasis on techniques to reduce anxiety. Over the 12-week period of the intervention, participants learn techniques for stress reduction that can be self-administered, such that the benefits of participation outlive the active period of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* MS Diagnosis
* 18 years or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of completion | Up to 12 weeks
  Acceptable rate is defined as at least 66% of participants who complete follow-up surveys.
Rate of adherence | Up to 12 weeks
  Acceptable rate is defined as at least 66% of sessions being attended.

SECONDARY OUTCOMES:
Score on the State Trait Anxiety Inventory (STAI) | Up to 12 weeks
  The STAI is a commonly used measure of trait and state anxiety that is scored from 20 (minimum score) to 80 (maximum score), with a higher scores indicating higher anxiety (worse outcome).

OTHER OUTCOMES:
Score on the Personal Health Questionnaire Depression Scale (PHQ-8) | Up to 12 weeks
  Mood as measured by change in depression or depressive symptoms will be measured with the 8-item PHQ-8 which is scored from 0 (minimum score) to 24 (maximum score), in which higher scores indicate higher depression or depressive symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Leavitt, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No